CLINICAL TRIAL: NCT07228481
Title: Randomised Controlled Trial of Two Different Cumulative Dosages of Roaccutane for Cystic Acne
Brief Title: Study of Two Dosages of Roaccutane in Cystic Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Premier Specialists, Australia (Other)
Collaborators: Roche Products Limited (Unknown)
Responsible Party: Principal Investigator, Dedee Murrell, Professor, Director of Premier Specialists, Premier Specialists, Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROC-ACNE
Record Dates: First submitted 2025-11-07; First posted 2025-11-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acne Cystic
MeSH Terms: interventions — Isotretinoin

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two treatment groups receiving different cumulative doses of Roaccutane (120 mg/kg or 150 mg/kg). Outcome assessments were performed by blinded evaluators.
Who Masked: Outcomes Assessor

ARMS (2):
- Roaccutane 120 mg/kg Group (Experimental): Participants in this arm received a cumulative dose of approximately 120 mg/kg of Roaccutane (isotretinoin) administered over the treatment period. Dosing was adjusted according to body weight and clinical response, following standard isotretinoin treatment protocols. The outcomes in this group were compared with those in the 150 mg/kg group to assess differences in efficacy, relapse rate, and adverse effects.
  Interventions: Drug: isotretinoin (Roaccutane)
- Roaccutane 150 mg/kg Group (Experimental): Participants in this arm received a cumulative dose of approximately 150 mg/kg of Roaccutane (isotretinoin) administered over the treatment period. Dosing was adjusted according to body weight and standard clinical guidelines for isotretinoin therapy. The outcomes for this group were compared with those of the 120 mg/kg group to evaluate differences in efficacy, relapse rates, and adverse effects.
  Interventions: Drug: isotretinoin (Roaccutane)

INTERVENTIONS:
Drug: isotretinoin (Roaccutane) — Oral administration of isotretinoin (Roaccutane) in capsule form, with cumulative dosage of 120 mg/kg. Dosing was adjusted according to body weight and administered over a period consistent with standard clinical protocols. The intervention was conducted as part of a randomized, single-blind controlled trial with blinded outcome assessment evaluating efficacy, relapse rates, and adverse events in patients with cystic acne.
  Arms: Roaccutane 120 mg/kg Group
Drug: isotretinoin (Roaccutane) — Oral administration of isotretinoin (Roaccutane) in capsule form, with cumulative dosage of 150 mg/kg. Dosing was adjusted according to body weight and administered over a period consistent with standard clinical protocols. The intervention was conducted as part of a randomized, single-blind controlled trial with blinded outcome assessment evaluating efficacy, relapse rates, and adverse events in patients with cystic acne.
  Arms: Roaccutane 150 mg/kg Group

SUMMARY:
This randomized, single-blind, controlled trial was initiated in 2001 to compare two cumulative isotretinoin doses (120 mg/kg vs 150 mg/kg) in patients with moderate-to-severe nodulo-cystic acne. Participants were assigned to receive a cumulative dose of either 120 mg/kg or 150 mg/kg, administered according to body weight and clinical response.

The primary objectives were to evaluate changes in total acne lesion counts and global acne severity grade from baseline through mid-treatment and end of treatment. Secondary objectives included assessing acne recurrence within 12 months after treatment completion and evaluating changes in acne scarring on the face, chest, and back over follow-up.

A small post-hoc extension cohort included patients who had not achieved satisfactory improvement after reaching their assigned cumulative dose and continued isotretinoin beyond standard targets. These patients were analysed descriptively.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects, of any age and any race
* Clinical diagnosis of nodulo-cystic acne as well as patients who have been unresponsive to standard acne vulgaris treatments

Exclusion Criteria:

* Pregnant or lactating female patients
* Female patients with polycystic ovarian syndrome, insulin resistance syndrome, previous use of Roaccutane, patients with congenital adrenal hyperplasia, patients with any internal malignancy (excluding skin cancer)
* Females of reproductive potential who refuse to take the oral contraceptive pill to take Roaccutane; patients who in the investigator's opinion would be unlikely to be compliant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2001-06-26 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Change in Total Acne Lesion Count During Isotretinoin Treatment | Baseline, Week 16, and end of treatment (defined as the visit at which the assigned cumulative dose of 120 mg/kg or 150 mg/kg was reached)
  Change in the total number of acne lesions (whiteheads, blackheads, papules, pustules, nodules, and deep pustules) measured on the face, chest, and back from baseline to week 16, and to the cumulative doses of 120 mg/kg and 150 mg/kg isotretinoin (Roaccutane).
  Results will be reported as the mean number of lesions at each time point. Lower counts indicate better clinical response.
Change in Acne Severity Grade During Isotretinoin Treatment | Baseline, Week 16, and end of treatment (defined as the visit at which the assigned cumulative dose of 120 mg/kg or 150 mg/kg was reached)
  Change in acne severity grade, ranging from 1 (least severe) to 8 (most severe), according to the classification described in Dermatology 1999;198:278-283 (Karger).
  Assessments are performed at baseline, week 16, and at cumulative isotretinoin doses of 120 mg/kg and 150 mg/kg.
  Results will be reported as mean acne grade (1-8 scale); lower scores indicate better outcome.

SECONDARY OUTCOMES:
Rate of Acne Relapse at 3 Months After End of Treatment | 3 months after completion of isotretinoin treatment
  Proportion of participants experiencing recurrence of inflammatory acne lesions requiring further systemic or topical therapy within 3 months following completion of isotretinoin treatment (at either 120 mg/kg or 150 mg/kg cumulative dose).
  Results will be expressed as percentage of participants with relapse.
Rate of Acne Relapse at 12 Months After End of Treatment | 12 months after completion of isotretinoin treatment
  Proportion of participants experiencing recurrence of inflammatory acne lesions requiring further systemic or topical therapy within 12 months following completion of isotretinoin treatment (at either 120 mg/kg or 150 mg/kg cumulative dose).
  Results will be expressed as percentage of participants with relapse.
Change in Acne Scarring Over Time | Baseline, end of treatment (defined as the visit at which the assigned cumulative dose of 120 mg/kg or 150 mg/kg was reached) and 12 months after completion of treatment
  Change in the number of atrophic and hypertrophic scars on the face, chest, and back from baseline to end of treatment and to 12-month follow-up. Results will be reported as mean scar counts at each time point.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study was conducted before data sharing requirements were established, and participants did not provide consent for their data to be publicly released. No data-sharing infrastructure or plan was created at the time of the study.

DOCUMENTS (3):
  • Study Protocol (2005-06-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT07228481/Prot_000.pdf
  • Informed Consent Form: For Minors (2000-10-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT07228481/ICF_001.pdf
  • Informed Consent Form: For Adults (2000-10-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT07228481/ICF_002.pdf